CLINICAL TRIAL: NCT06972069
Title: Tolerance Through Mixed Chimerism (Sip-Tego)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tatsuo Kawai, MD, PhD (Other)
Collaborators: Eledon Pharmaceuticals (Industry); ITB-Med LLC (Industry)
Responsible Party: Sponsor-Investigator, Tatsuo Kawai, MD, PhD, Physician, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000818
Record Dates: First submitted 2025-04-22; First posted 2025-05-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Kidney Failure; Transplant Recipient (Kidney); Transplant Tolerance; Immunosuppresion; Immunosuppression After Kidney Transplantation
Keywords: Tolerance; Transplant without immunosuppression; kidney transplant
MeSH Terms: conditions — Renal Insufficiency | interventions — Transplantation Conditioning; Rituximab; siplizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recipient (Experimental): Recipient of kidney and bone marrow transplant
  Interventions: Procedure: Combined Kidney/Bone Marrow Transplant; Drug: Conditioning Regimen (Rituxan, Siplizumab, Cyclophosphamide, Tegoprubart)
- Donor (Other): Living donors of kidney and bone marrow transplant
  Interventions: Procedure: Donation of Kidney / Bone Marrow

INTERVENTIONS:
Procedure: Combined Kidney/Bone Marrow Transplant — The conditioning regimen to be used in this protocol consists of an ordered series of procedures and treatments including thymic irradiation, low-dose cyclophosphamide, antibody administration (Siplizumab, rituximab and tegoprubart), and bone marrow cell infusion.
  Arms: Recipient
Procedure: Donation of Kidney / Bone Marrow — The donor will undergo nephrectomy and under general anesthesia. Donors will undergo bone marrow harvested under general anesthesia. Sufficient marrow will be obtained to provide at least 2 x 108 nucleated cells per kilogram weight of the recipient.
  Arms: Donor
Drug: Conditioning Regimen (Rituxan, Siplizumab, Cyclophosphamide, Tegoprubart) — Recipients will receive a conditioning regimen that includes rituximab on study day -6 and -2, Siplizumab (0.6mg/kg) on day -6, -1, 0 and +1, cyclophosphamide (CP, 22.5mg/kg) on days -5 and -4. Tegoprubart (Fc-modified anti-CD154 mAB, Eledon Pharm) 20mg/kg will be administered on days 0, 2, 5, 12 and 19).
  Arms: Recipient

SUMMARY:
This is an open-label, single-institution study to assess the safety and the efficacy of the Sip-Tego regimen for the induction of donor-specific immunologic unresponsiveness to a renal allograft. The investigators propose to treat 6 adult subjects in end-stage renal disease (ESRD) who do not demonstrate evidence of prior sensitization.

DETAILED DESCRIPTION:
The conditioning regimen to be used in this protocol consists of an ordered series of procedures and treatments including thymic irradiation, low-dose cyclophosphamide, antibody administration (Siplizumab, rituximab and tegoprubart), and bone marrow cell infusion. The surgical techniques for the renal transplant will be accomplished according to the surgeon's clinical judgment and experience using standard techniques in use at the institution. The donor nephrectomy will be accomplished according to the surgeon's clinical judgment and experience. The conditioning regimen requires six days leading up to the day of transplantation, which is designated as study Day 0. Negative numbers in descending order designate days pre-transplant, while positive numbers in ascending order designate days post-transplant. Refer to Figure 2 in Section 1.2. for the schema of the conditioning regimen.

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Male or female 18-65 years of age.
2. Subjects with chronic kidney disease stage V (GFR<15ml/min/1.73m2) or ESRD who are treated or imminently be treated with either hemodialysis or peritoneal dialysis.
3. Candidate for a living-donor renal allograft from an HLA matched or mismatched donor
4. First or second renal transplant.
5. EBV Seropositive
6. Use of FDA-approved methods of contraception by all recipients from the time that study treatment begins until 104 weeks (24 months) after renal transplantation
7. Ability to understand and provide informed consent.
8. Negative COVID-19 test during screening and two days prior to procedure

Recipient Exclusion Criteria:

1. ABO blood group-incompatible renal allograft
2. Participant with a donor-specific antibody (DSA) within 6 months prior to transplant
3. Persistent Leukopenia (WBC less than 2,000/mm3) or thrombocytopenia (<100,000/mm3)
4. Seropositivity for HIV-1, hepatitis B core antigen, or hepatitis C virus (confirmed by hepatitis C virus RNA); or positivity for hepatitis B surface antigen.
5. Untreated Infection
6. Left ventricular ejection fraction < 40% as determined by TTE or clinical evidence of heart failure.
7. Forced expiratory volume FEV1 or DLCO < 50% of predicted.
8. Lactation or pregnancy.
9. Patients with active cancer or those with a high risk of recurrence following the American Transplant Society
10. Underlying renal disease etiology with a high risk of disease recurrence in the transplanted kidney (such as non-genetic primary focal segmental glomerulosclerosis dense deposit disease, C3 glomerulonephritis, and, atypical hemolytic uremic syndrome).
11. Prior dose-limiting radiation therapy for treatment of malignant disease.
12. Known genetic disease or family history that may result in greater sensitivity to the effects of irradiation, or a physical deformity that would preclude adequate shielding or appropriate dosing during the irradiation component of the conditioning regimen. This includes long term cigarette smoking or a family history of malignancy.
13. Enrollment in other investigational drug studies within 30 days prior to enrollment.
14. Abnormal (>2 times lab normal) values for (a) liver function chemistries (ALT, AST, AP), (b) bilirubin, (c) coagulation studies (PT, PTT) , or any patients on chronic anticoagulation therapy.
15. Allergy or sensitivity to any component of Cyclophosphamide, tacrolimus, Siplizumab, Tegoprubart, or rituximab.
16. The presence of any medical condition that the investigator deems incompatible with participation in the trial. This includes a history of alcohol abuse or illicit drug use/dependence.
17. Any chronic or intermittent administration of immunosuppressant medication (such as for inflammatory bowel disease or asthma)
18. Subjects who have non-insulin dependent diabetes (NIDDM) without good blood glucose control (HbA1c<8%). Subjects with severe diabetes-related complications, such as advanced retinopathy, gastroparesis, or severe neuropathy that significantly impair their ability to perform normal, independent daily activities, will also be excluded.

Donor Inclusion Criteria:

1. Male or female 18-70 years of age.
2. For females of childbearing potential: a serum pregnancy test showing negative results.
3. Excellent health per conventional pre-donor workup (medical and psychosocial evaluation)
4. Acceptable laboratory parameters (hematology in normal or near-normal range; Liver function <2 times the upper limit of normal, and normal creatinine).
5. Negative for viral infection with HBV (HbsAg and NAT), HIV (antibody and NAT), HCV (NAT), or HTLV-1.
6. Cardiac/pulmonary function within normal limits (CXR, ECG).
7. Ability to understand and provide informed consent.
8. Meets standard institutional criteria for bone marrow aspiration and kidney donation.
9. Negative COVID-19 test during screening and two days prior to procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Induction of mixed chimerism without chimeric transition syndrome | 7 Years
  This will be measured by a chimerism level of >0% donor chimerism at anytime post transplant, and when the level is returning to 0% chimerism there is no evidence of chimeric transition syndrome. This is defined in the protocol by any of the following The clinical symptoms of CTS include acute kidney injury with rapid deterioration of kidney function (elevated creatinine, decreased blood flow to the renal allograft by US), minor to moderate fever, fluid retention or peripheral edema.
Achievement of IS minimization (tacrolimus or Belatacept monotherapy) | 7 Years
  This will be measured by a patient weaning and maintaining only one agent of immunosuppression (either Tacrolimus or Belatacept)
Number of patients who complete full immunosuppression withdrawal | 7 Years
  The number (and therefore percentage) of patients who discontinue all immunosuppression (ie. completely stop Tacrolimus or Belatacept)

SECONDARY OUTCOMES:
Participants who are alive at the end of the study | 7 Years
Kidney Graft Survival | 7 Years
Incidence of CTS | 7 Years
Incidence of Acute Rejection | 7 Years
Incidence of Donor Specific Antibody development | 7 Years
Incidence of Chronic Rejection | 7 Years
Incidence of GVHD (Acute or Chronic) | 100 days
Incidence of clinically significant or resistant Opportunistic Infections | 7 Years
Recovery of neutrophils to normal range | 7 Years
  A neutrophil count that is within normal lab range (after early myelosuppression from conditioning regimen)
Recovery of Platelets to normal range | 7 Years
  A Platelet count that is within normal lab range (after early myelosuppression from conditioning regimen)
Incidence of Serious Adverse Events | 7 Years
Incidence of Radiation related toxicities | 7 Years

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuo Kawai, MD PhD, Principal Investigator — Principal Investigator / Transplant Surgeon
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.massgeneral.org/transplant/transplant-programs/tolerance